CLINICAL TRIAL: NCT00723944
Title: A Prospective, Randomized-controlled Multicenter Study of the Osseotite Certain Lateralized Implanting Short-span Fixed Bridge Cases for Preservation of Crestal Bone
Brief Title: A Study of the Performance of Certain Prevail Implants Used in Short Fixed Cases
Acronym: RadioCity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2302
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: dental implants; Osseotite Certain Prevail; Lateralized; non-lateralized; Osseotite Certain; multicenter; randomized; clinical study; partial edentulism; single stage; early loading; crestal bone level; short fixed bridge
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Osseotite Certain Prevail (Active Comparator): Dental implant with lateralized design
  Interventions: Device: Osseotite Certain Prevail
- Osseotite Certain (Placebo Comparator): Dental implant without the lateralized design
  Interventions: Device: Osseotite Certain

INTERVENTIONS:
Device: Osseotite Certain Prevail — Root form titanium dental implant
  Other Names: Osseotite; Certain; Prevail
  Arms: Osseotite Certain Prevail
Device: Osseotite Certain — Dental implant without the lateralized design
  Other Names: Osseotite; Certain
  Arms: Osseotite Certain

SUMMARY:
This prospective, randomized study evaluates the performance and crestal bone changes difference between the Osseotite Certain Prevail vs the non-lateralized design of the implant.

Study (null) hypothesis: the crestal bone changes that take place after placement and loading of the Osseotite lateralized implants will be the same as for similar but non-lateralized Osseotite Certain implants.

DETAILED DESCRIPTION:
This is a prospective, randomized-controlled study where patients with qualifying partial edentulism received a short fixed bridge restoration. Each implant site was randomized to receive either the test (Osseotite Certain Prevail) or the control non lateralized version of the Osseotite Certain implant. All implants were placed in a single-stage manner with temporary provisionalization taking place two months after implant placement. Enrollment continued until 10 patients (approximately 30 implants) were treated at each participating study center.

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and any race greater than 18 years of age
* patients for whom a decision has already been made to use dental implants for treating an existing dental condition specifically: a partially edentulous short fixed case of less than 4 implants in the maxilla or mandible; no cantilevers are allowed, but one interior crown may be a pontic
* patients must be physically able to tolerate conventional surgical and restorative procedures
* patients must agree to be evaluated for each study visit, especially the yearly follow-up visit

Exclusion Criteria:

* patients with active infection or severe inflammation in the areas intended for the implants
* patients with more than 10 cigarette per day smoking habit
* patients with uncontrolled diabetes mellitus
* patients with metabolic bone disease
* patients who have had treatment with therapeutic radiation to the head within the past 12 months
* patients in need of allogenic bone grafting at the site of the intended study implant
* patients who are pregnant at the screening visit
* patients with evidence of severe para-functional habits such as bruxing or clenching
* patients with cantilevers and more than one pontic per bridge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2005-02; Primary Completion 2007-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anton Friedmann, DMD, Principal Investigator — Charite- Zentrum fur Zahnmedizin
Locations (1):
- Charite- Universitatsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A minimum of 100 patients were enrolled across all participating centers, with enrollment beginning in January 2005. Enrollment period remained open until April 2006. Three participating sites were Universities and seven were private practices.
Pre-assignment Details: Pre-treatment included a screening visit (enroll those meeting all inclusion criteria), signing informed consent, and pre-surgical data collection.Patients returned for implant placement surgery, followed by temporary prosthesis placement at 2 months.
Groups:
- Osseotite Certain Prevail Implant: Patients with dental implant with internal connection and expanded, lateralized design at coronal portion
- Osseotite Certain Implant: Patients with dental implant with internal connection and without the expanded, lateralized design at coronal portion
Period: Implant Placement Surgery
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Started | 52 (number of individual implant units is 148) | 50 (number of individual implant units is 138)
Completed | 52 (number of individual implant units completing is 148) | 50 (number of individual implant units completing is 138)
Not Completed | 0 | 0
Period: Permanent Prosthesis Placement
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Started | 52 (number of individual implant units is 148) | 50 (number of individual implant units is 138)
Completed | 49 (number of individual implant units completing is 134) | 41 (number of individual implant units completing is 112)
Not Completed | 3 | 9
Not completed — Adverse Event | 1 | 7
Not completed — Lost to Follow-up | 2 | 2
Period: One Year Post Placement Follow-up
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Started | 49 (number of individual implant units is 134) | 41 (number of individual implant units is 112)
Completed | 48 (number of individual implant units completing is 130) | 37 (number of individual implant units completing is 108)
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 4
Period: Two Year Post Placement Follow-up
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Started | 48 (number of individual implant units is 130) | 37 (number of individual implant units is 108)
Completed | 48 (number of individual implant units completing is 130) | 37 (number of individual implant units completing is 108)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 38 | 78
  >=65 years | 12 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 31 | 31 | 62
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
  Italy | 19 | 17 | 36
  France | 6 | 5 | 11
  Germany | 8 | 8 | 16
  Sweden | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Crestal Bone Regression (Amount of Bone Measured) Around Each Implant Unit
Description: Millimeters of crestal bone observed and measured in a radiograph of each study implant is measured and averaged to obtain the mean crestal bone loss or gain for each implant unit.
Time Frame: 1 year
Population: population represents all patients receiving test and control implants enrolled in the study, but only those implants achieving integration (lack of mobility) were analyzed and reported here up to the 12 months follow-up stage.
Measure: Mean (Standard Error); unit: millimeters
Units Other Than Participants: implants
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Number analyzed (Participants) | 48 | 37
Number analyzed (implants) | 130 | 108
millimeters | -0.7705 (0.1567) | -0.6648 (.1158)

2. Secondary Outcome: Osseous Integration
Time Frame: 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event reporting is collected from day of the study to present, currently 4 years study duration.
Description: Adverse event data is collected by patient questionaire and visual inspection (assessment) of patient's mouth during each study event visit.
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50
Other Adverse Events (participants affected / at risk) | 4/52 | 19/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osseotite Certain Prevail Implant (N=52) | Osseotite Certain Implant (N=50)
Loss of implant integration (Surgical and medical procedures) | 4 (4) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall furnish SPONSOR with a copy of any proposed publication thirty (30) days prior to submission for publication for review and comment. SPONSOR may request PI to delay publishing such proposed publication for a maximum of an additional sixty (60) days in order to protect the potential patentability of any invention described therein.